CLINICAL TRIAL: NCT02494258
Title: A Phase 2, Open-Label, Single-Arm Rollover Study to Evaluate Long-Term Safety in Subjects Who Participated in Other Celgene Sponsored CC-486 (Oral Azacitidine) Clinical Trials in Hematological Disorders
Brief Title: A Study to Evaluate Long-term Safety of CC-486 (Oral Azacitidine) in Subjects With Hematological Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-GEN-001; 2023-503272-25 (EudraCT Number)
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Neoplasm; Neoplasms; Hematologic Malignancies
Keywords: CC-486; Oral Azacitidine; hematological disorders; rollover study; open label; Onureg
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Hematologic Diseases | interventions — cc-486; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Azacitidine (CC-486) (Experimental): This study is an open-label, single-arm study and is divided into the screening period, treatment period and follow-up period. It is intended to evaluate the long-term safety of CC-486 and is to be taken at the same dose, schedule and frequency used from the last dose of CC-486 given in the parent study.
  Interventions: Drug: CC-486

INTERVENTIONS:
Drug: CC-486 — The subject will continue at the same dose, frequency and schedule used for the last dose of CC-486 given in the preceding CC-486 study. Subjects are allowed to rollover after the last cycle is finished and before the new cycle begins in the parent protocol. There is a 7 day window from End of Study on the parent protocol and when the participant will start Day 1 of the rollover study.
  Other Names: Oral Azacitidine; BMS-986345; Onureg

SUMMARY:
Rollover study supporting hematological disorder indications from Celgene sponsored CC-486 (oral azacitidine) protocols eligible for participation in the study.

DETAILED DESCRIPTION:
The open-label, multicenter, multinational rollover study is intended to evaluate the safety of CC-486 (oral azacitidine), while providing continued treatment with CC-486 for subjects who are receiving single agent CC-486 at the time of transition to the rollover study and tolerated the protocol prescribed regimen in Celgene-sponsored trials, and whom in the opinion of the Investigator may derive clinical benefit from continuing treatment with CC-486. Subjects' survival will also be followed if required by the parent CC-486 study protocol. If approved by Celgene, subjects from any ongoing or future Celgene sponsored CC-486 studies in hematological disorders will be included in this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Previously participated in, and received oral azacitidine, and continues to fulfill the eligibility criteria in one of the parent oral azacitidine clinical trials.

   The Investigator believes the subject is tolerating treatment with oral azacitidine monotherapy and continued oral azacitidine treatment is of benefit to the subject.
2. Understand and voluntarily sign an informed consent document prior to any study related assessments or procedures being conducted.
3. Willing and able to adhere to the study visit schedule and other protocol requirements.
4. Females of childbearing potential (FCBP) may participate, provided that the participant meets the following conditions:

   1. Have two negative pregnancy tests as verified by the Investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.
   2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with highly effective contraception without interruption, during screening, during the study treatment (including dose interruptions), and for 6 months after discontinuation of study treatment, or longer if required for each compound and/or by local regulations.

Subjects must satisfy the following criteria to participate in the Survival Follow-up phase:

1. In order to be enrolled for the survival follow-up in the Follow-up Phase of the rollover study, subjects must have been in a parent oral azacitidine study where monitoring for survival was required and have signed informed consent for follow-up phase.
2. Understand and voluntarily sign an informed consent document for this study.
3. Willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from receiving investigational product in the study:

1. Concomitant use of drugs that are prohibited.
2. Prior chemotherapy (including injectable azacitidine) or radiotherapy or any investigational agent after the last dose of oral azacitidine administered as part of the parent oral azacitidine study.
3. Subjects have met one or more criteria for discontinuation as stipulated in the parent oral azacitidine study.
4. Subjects received oral azacitidine in combination with another compound during a parent oral azacitidine study (Subjects form multi-arm parent oral azacitidine studies will be allowed to enroll into the rollover study, if the subject is receiving single-agent oral azacitidine at the time of transition into the rollover study).
5. A subject's transition into rollover study ≥ 45 days after End of the Study visit of the parent oral azacitidine study
6. Pregnant or lactating females.

There are no exclusion criteria to prevent entry or remaining on the follow-up phase of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Approximately 5 years
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health including laboratory test values, regardless of etiology.

SECONDARY OUTCOMES:
Overall Survival | Up to 5 years
  Time from randomization until death from any cause.
  If required by the parent CC-486 study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (3):
  - Local Institution - 101, Gainesville, Florida
  - Local Institution - 103, Baltimore, Maryland
  - Local Institution - 102, Houston, Texas
- Manchester Royal Infirmary, Manchester, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com